CLINICAL TRIAL: NCT06419764
Title: Combining Chinese Medicine and Nutrition to Enhance Weight Loss After Bariatric Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Hua Meng, Director of the General Surgery Department & Obesity and Metabolic Disease Center of China-Japan Friendship Hospital, China-Japan Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCMNEWLABS
Record Dates: First submitted 2024-05-14; First posted 2024-05-17 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Traditional Chinese Medicine Treatment; Weight Change
MeSH Terms: conditions — Body Weight Changes | interventions — Diet

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nutrition intervention group (Active Comparator): Postoperative patients are routinely provided with meal replacement recommendations and dietary plans.
  Interventions: Other: Diet and meal replacements
- Traditional Chinese Medicine combined with nutritional intervention (Experimental): Chinese herbal treatment is given on the basis of routine dietary intervention.
  Interventions: Drug: Spleen Invigorating and Weight Reducing Decoction; Other: Diet and meal replacements

INTERVENTIONS:
Drug: Spleen Invigorating and Weight Reducing Decoction — Composition: Raw Astragalus (Huang Qi) 5g, Cang Zhu 5g, Fructus Aurantii Immaturus (Zhi Shi) 3g, Prepared Rhubarb (Shu Jun) 3g, Red Peony Root (Chi Shao Yao) 3g, Crataegus (Shan Zha) 3g, Tribulus (Bai Jie Li) 2g, Cimicifuga (Sheng Ma) 1g.
  Granule form, for oral administration. Take 1 dose daily (2 bags, once in the morning and once in the evening, dissolved in water), for a course of 1 month.
  Arms: Traditional Chinese Medicine combined with nutritional intervention
Other: Diet and meal replacements — The dietitian provides recommended meal plans based on body weight, and meal replacements are used postoperatively.

SUMMARY:
This study aims to investigate the effects of Chinese herbal granule preparations on improving gastrointestinal symptoms in patients after bariatric surgery. It seeks to establish a novel treatment model that combines bariatric surgery with traditional Chinese medicine, providing clinical practice with additional evidence-based medical support.

ELIGIBILITY:
Inclusion Criteria:

1. BMI ≥ 27.5 kg/m²;
2. Undergoing metabolic bariatric surgery;
3. Traditional Chinese Medicine syndrome differentiation classified as Spleen Deficiency and Excess Dampness syndrome.

Exclusion Criteria:

1. Contraindications for metabolic bariatric surgery;
2. Type 1 diabetes;
3. Complicated by other significant systemic diseases, such as severe liver and kidney diseases, malignant tumors, psychiatric disorders, etc;
4. Concurrent use of other medications or treatments that may affect body weight, such as metformin, semaglutide, endoscopic interventions, etc;
5. Pregnant or lactating women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Percentage change in body weight | Before bariatric surgery, 1 month after surgery, and 3 months after surgery.

SECONDARY OUTCOMES:
Traditional Chinese Medicine syndrome score | Before bariatric surgery, 1 month after surgery, and 3 months after surgery.
blood glucose indicators | Before bariatric surgery, 1 month after surgery, and 3 months after surgery.
  HbA1c, blood glucose, insulin levels
blood lipid profile | Before bariatric surgery, 1 month after surgery, and 3 months after surgery.
  total cholesterol, triglycerides, high-density lipoprotein cholesterol, low-density lipoprotein cholesterol

CONTACTS AND LOCATIONS:
Locations (1):
- China-Japan Friendship Hospital, Beijing, China